CLINICAL TRIAL: NCT03214068
Title: Evaluation of the Pattern of Thyroid Dysfunctions in Patients With Metabolic Syndrome
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, GAAbdelhay, Resident doctor of internal medicine, Assiut University
Other Study IDs: 17100051
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study on evaluation the pattern of TD in MetS population may help us to know the magnitude of overlap of these two disease entities and may highlight the importance of thyroid function tests in patients with MetS. This can lead to proper planning and adequate management strategies, resulting in significant reduction in cardiovascular morbidity and mortality due to MetS with TD. Thus, this study aims to evaluate the pattern of TD in patients with MetS and to explore the relationship between TD and components of the MetS.

DETAILED DESCRIPTION:
The metabolic syndrome (MetS) is a clustering of multiple risk factors for atherosclerotic cardiovascular disease such as central obesity, impaired fasting glucose (IFG) or type 2 diabetes mellitus (T2DM), elevated triglyceride (TG), reduced high density lipoprotein cholesterol (HDL-C) and hypertension (HTN).This cluster of metabolic abnormalities is associated with increased risk for atherosclerotic cardiovascular disease and type 2 diabetes mellitus Despite of the controversy on its definition, it is estimated that one out of four people around the world suffers from MetS. The prevalence of MetS is increasing all over the world.

Thyroid hormones play an important role in regulating energy homeostasis, carbohydrate, lipids and protein metabolism. These hormones accelerate metabolic processes and may be associated with metabolic syndrome. Hyperthyroidism is usually associated with low cholesterol and glucose intolerance; whereas hypothyroidism is associated with high cholesterol tendency, and patients are prone to weight gain and cardiac signs like bradycardia. Thyroid functions affect the components of MetS including HDLcholesterol (HDL-C), triglycerides (TG), blood pressure and plasma glucose.

Thyroid dysfunction (TD) is defined as the altered serum thyroid stimulating hormone (TSH) level with normal or altered thyroid hormones (free triiodothyronine and free thyroxine.TD is risk factors for CardioVascular Disease mediated by the effects of thyroid hormones on lipid and glucose metabolism and blood pressure, hence on components of MetS.MetS and TD are both characterized by a cluster of common abnormalities such as abdominal obesity, hyperglycemia, HTN, reduced HDL-C, and elevated TG and recognized independent risk factors of ASCVD ..Thyroid dysfunction, prominently subclinical hypothyroidism has been observed more frequently in metabolic syndrome patients than general population .

The study on evaluation the pattern of TD in MetS population may help us to know the magnitude of overlap of these two disease entities and may highlight the importance of thyroid function tests in patients with MetS. This can lead to proper planning and adequate management strategies, resulting in significant reduction in cardiovascular morbidity and mortality due to MetS with TD. Thus, this study aims to evaluate the pattern of TD in patients with MetS and to explore the relationship between TD and components of the MetS.

ELIGIBILITY:
Inclusion Criteria:

* Patients satisfying the 2005 Revised National Cholesterol Education Program/AdenosineTri Phosphate III which have three out of five of the following criteria:

  1. Central obesity - defined as waist circumference ≥102 cm for Men and ≥88cm for women.
  2. Raised triglycerides: ≥ 150 mg/dL, or specific treatment for this lipid abnormality.
  3. Reduced HDL cholesterol: < 40 mg/dL in males,< 50 mg/dL in females, or specific treatment for this lipid abnormality
  4. Raised blood pressure: systolic BP ≥130 or diastolic BP ≥85 mm Hg, or treatment of previously diagnosed hypertension.
  5. Raised fasting plasma glucose :( FPG) ≥100 mg /dL, or previously diagnosed type 2 diabetes.

     * knownly diagnosed diabetes mellitus .
     * hypertension diagnosed patients .
     * obese patients.

Exclusion Criteria: 1. Known hypothyroid or sub-clinical hypothyroid or hyperthyroid patients or on treatment.

2. Patients with liver disorders, renal disorders, congestive cardiac failure, pregnant women.

3. Patients with history of respiratory disease, malignancy, Smokers, alcoholics, 4. patients receiving medication that may alter thyroid functions or lipid levels,

-

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include 100 patients with metabolic syndrome (MetS) who fulfilled criteria according to the 2005 Revised National Cholesterol Education Program/ATP III. Age and sex matched100 healthy persons who have no features of metabolic syndrome will be included in the study as a control group .
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
Thyroid stimulating hormone | 2 years.
  Evaluation of thyroid dysfunctions in patients with metabolic syndrome

SECONDARY OUTCOMES:
Lipid profile | 2 years
  To evaluate the associations between thyroid hormones levels and components of metabolic syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Udenze I, Nnaji I, Oshodi T. Thyroid function in adult Nigerians with metabolic syndrome. Pan Afr Med J. 2014 Aug 29;18:352. doi: 10.11604/pamj.2014.18.352.4551. eCollection 2014. PMID 25574328
- See also: Thyroid function in adult Nigerians with metabolic syndrome — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4282811/
- Available data/document: Clinical Study Report — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4282811/